CLINICAL TRIAL: NCT00175838
Title: A Randomised Trial to Compare Aspirin vs Hydroxyurea/Aspirin in 'Intermediate Risk' Primary Thrombocythaemia and Aspirin Only With Observation in 'Low Risk'Primary Thrombocythaemia
Brief Title: Primary Thrombocythaemia 1 Trial
Acronym: PT-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Principal Investigator, Anthony Green, Professor of Haemato-Oncology, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A05033; EUdraCT no:2004-000245-38; ISRCTN: 72251782
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Thrombocythemia; Myeloproliferative Disorder
Keywords: Primary Thrombocythmeia; Hydroxyurea; Randomised; Thrombosis; Haemorrhage
MeSH Terms: conditions — Thrombocytosis; Myeloproliferative Disorders; Thrombosis; Hemorrhage | interventions — Hydroxyurea; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intermediate risk group (Active Comparator): Intermediate risk patients are randomised to a either a group receiving Aspirin only, or a group receiving both Hydroxyurea and Aspirin.
  Interventions: Drug: Hydroxyurea; Drug: Aspirin
- Low risk group (Active Comparator): Patients are given Aspirin only with observation.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Hydroxyurea — Hydroxyurea (or hydroxycarbamide) is an antineoplastic drug commonly used to treat haematological malignancies.
  Other Names: Hydroxycarbamide
  Arms: Intermediate risk group
Drug: Aspirin — Aspirin is an anti-aggregating agent, and has been shown to reduce/alleviate minor ischaemic symptoms.

SUMMARY:
The purpose of this trial is to see if Hydroxyurea + aspirin is a better treatment than aspirin alone for Intermediate Risk Primary Thrombocythemia (PT) patients.

DETAILED DESCRIPTION:
The myeloproliferative disease, primary thrombocythaemia (PT), has a median age of presentation of 60 years but is increasingly being recognised at an earlier age. The risks of the untreated condition are micro-vascular and major vessel occlusive events and haemorrhage. Older patients and those with a previous thrombosis are particularly prone to experience a significant vascular occlusive event. An anti-aggregating agent, such as aspirin, has been shown to reduce/alleviate minor ischaemic symptoms. Therefore, except in patients with haemorrhagic symptoms, peptic ulceration and known side-effects to aspirin, the use of low-dose aspirin is appropriate.

Myelofibrotic and acute leukaemic transformations can be long-term complications of PT. The ability of therapeutic agents to delay myelofibrosis or reduce/increase the incidence of acute leukaemia in prospective studies is unknown. However, examination of retrospective data provides anxiety about the leukaemogenic risk of the commonly used cytoreductive agent, hydroxyurea. From an analysis of a few relatively small studies of primary thrombocythaemia, the incidence of acute leukaemic transformation in selected patients treated with hydroxyurea has been given as 5-10% over 4-11 years (1).

Based on the risk factors for vascular occlusion, older patients with a thrombotic history and high platelet count can be separated into a 'high' risk group. There is evidence from a randomised prospective study of 'high-risk' patients that cytoreduction with hydroxyurea significantly reduces vascular occlusion (2). The observed reduction in this prospective study of 29 months median duration was from 24% for those not given cytoreductive treatment to 3.6% for those receiving hydroxyurea - approximately a six-fold reduction. In another prospective study where all patients received hydroxyurea, an incidence of major thrombotic events was 5.6%/year (3). In these high-risk patients, cytoreductive treatment should therefore be given. The high risk arm of the PT1 trial, which has now closed, assessed the cytoreductive treatment of choice for these high risk patients and the results suggest that hydroxyurea plus aspirin is superior to anagrelide plus aspirin (4).

In the patients at lower risk of vascular occlusion the dilemma is that the risk of vascular occlusion in untreated patients is relatively low, but includes major life-threatening events. In two small prospective studies of these patients not receiving platelet lowering agents, the observed major complications were 3% and 4.1% per year and the total complications were 5.1% and 10.5% per year respectively (1). Cyto-reductive treatment should prevent such events and one could predict a similar reduction in complications as seen in the high-risk patients. However, there is evidence that in patients under the age of 40 years the complication rate is only one quarter of that seen in patients aged 40 - 59 years (5). Therefore it has been decided to divide these patients at lower risk of vascular occlusion into 'intermediate' and 'low risk' groups. Patients aged 40-59 years will fall into the 'intermediate risk' group and will be randomised to cytoreduction or not, while all will receive aspirin. Patients under 40 years will form the 'low-risk' group and will receive aspirin alone. Cyto-reductive treatment might also delay myelofibrotic transformation as observed in primary polycythaemia. However, this benefit and the possible reduction in vaso-occlusive episodes need to be balanced against the potential long-term risk of increasing acute leukaemic transformation.

ELIGIBILITY:
Inclusion Criteria:

* The proposal is to include as many patients with PT as possible including previously diagnosed patients whether or not they have received treatment. Thus all patients are eligible assuming they meet the diagnostic criteria and they do not have any exclusion criterion (see below). It will be necessary to stratify patients according to their previous treatment. This information will be collected on entry to the study. Informed consent is of course required where there is a change of therapeutic strategy.

The diagnostic criteria for primary thrombocythaemia are:

* Platelet count > 600x109/l.
* No evidence of overt polycythaemia(confirmed by RCM if necessary)or of polycythaemia masked by co-existent iron deficiency.
* No Philadelphia chromosome.
* Absence of peripheral blood and/or marrow appearances of myelodysplasia, or myelofibrosis.
* No known cause of reactive thrombocytosis. Particular care should be taken to exclude iron deficiency in pre-menopausal women.

Notes:

* In asymptomatic patients, the platelet count should be observed for a period of at least 2 months to confirm >600x109/l, and to allow any cause of reactive thrombocytosis to become overt.
* If the PCV is above normal upper limit (that is, males >0.51, females >0.48) or in high normal range in a patient with palpable splenomegaly measure RCM. Iron deficient primary polycythaemia (polycythaemia vera) is strongly suggested if Hb/PCV is normal in the presence of iron deficient red cell changes. In this situation, iron therapy is potentially dangerous.
* Exceeding rarely, bcr-abl positive Philadelphia chromosome negative patients present with high platelet counts with little or no elevation in WBC count. The features that suggest it is necessary to examine for bcr-abl, are:- basophilia, left-shift in WBC, granulocyte count >16x109/l, difficulty in controlling platelet count, megakaryocytes of low ploidy (NAP is usually unhelpful).
* A normal ESR, CRP or plasma viscosity is useful in excluding a reactive thrombocytosis.
* Written informed consent obtained in accordance with NCRI requirements.
* Patients with impaired hepatic / renal function are not excluded although the respective biochemical tests should be monitored during therapy and reduced doses of cytoreductive agent should be used, particularly in the case of hydroxyurea and renal dysfunction.

Exclusion Criteria:

High risk features (any of the following):

* Age >or= 60 years
* Platelet count > or= 1500x109/l (current or previous) (a)
* History of ischaemia, thrombosis or embolic events (including erythromelalgia) (b)
* Haemorrhage considered to be related to PT (b)
* Presence of hypertension (c)or diabetes (d)
* The manufacturers of hydroxyurea state that it should be avoided in pregnancy and in lactating women. Similarly, hydroxyurea should not be prescribed for women when there is doubt about their use of an effective contraceptive method.
* Exclude patient from hydroxyurea therapy and, therefore, from the 'intermediate' risk randomisation if the patient has current leg ulcers.

Notes on the definition of high risk:

* In patients with borderline counts the allocation of a patient to a high risk group based on platelet count alone should rely on at least three samples taken on separate occasions over at least 2 months.
* Documentation of previous thrombo-embolic, ischaemic and haemorrhagic events should be given on the patient's entry proforma.
* Hypertension is defined as those patients requiring hypotensive therapy.
* Diabetes is defined as those patients requiring therapy with a hypoglycaemic agent.

Ages: 40 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1398 (Actual)
Dates: Start 1997-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Does hydroxyurea reduce thrombosis and major haemorrhage when added to aspirin? | 14 years
  Reducing thrombosis and major haemorrhage are specific key measurements in this group of patients for whom thrombotic events are very likely to occur.

SECONDARY OUTCOMES:
Does treatment modality alter the risk of leukaemic or myelofibrotic transformation? | 14 years

CONTACTS AND LOCATIONS:
Overall Officials: Anthony R Green, Prof, Study Director — Addenbrooke's Hospital and University of Cambridge; Claire Harrison, Dr, Principal Investigator — St Thomas' Hospital
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambs, United Kingdom

REFERENCES:
- [Derived] Godfrey AL, Campbell PJ, MacLean C, Buck G, Cook J, Temple J, Wilkins BS, Wheatley K, Nangalia J, Grinfeld J, McMullin MF, Forsyth C, Kiladjian JJ, Green AR, Harrison CN; United Kingdom Medical Research Council Primary Thrombocythemia-1 Study; United Kingdom National Cancer Research Institute Myeloproliferative Neoplasms Subgroup; French Intergroup of Myeloproliferative Neoplasms; the Australasian Leukaemia and Lymphoma Group.. Hydroxycarbamide Plus Aspirin Versus Aspirin Alone in Patients With Essential Thrombocythemia Age 40 to 59 Years Without High-Risk Features. J Clin Oncol. 2018 Dec 1;36(34):3361-3369. doi: 10.1200/JCO.2018.78.8414. Epub 2018 Aug 28. PMID 30153096